CLINICAL TRIAL: NCT04549493
Title: Effectiveness of Trauma Management Therapy and Prolonged Exposure Therapy for the Treatment of Post-Traumatic Stress Disorder in an Active Duty Sample: A Comparison Study
Brief Title: Effectiveness of Trauma Management Therapy and Prolonged Exposure Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH18C0331
Record Dates: First submitted 2020-05-22; First posted 2020-09-16 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-12

CONDITIONS: PTSD
Keywords: Trauma Management Therapy; Exposure Therapy; Group Therapy; PTSD; Military
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Implosive Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trauma Management Therapy (Active Comparator): 1. Trauma Management Therapy (TMT; Turner, Beidel, & Frueh, 2005): TMT is a multicomponent behavioral treatment program designed to target various aspects of chronic PTSD - reducing emotional and physiological reactivity to traumatic cues, reducing intrusive symptoms and avoidance behavior, improving interpersonal skills and emotion modulation (e.g., anger control), and increasing the range of enjoyable social activities. In this investigation and in line with our previous publications, TMT will include virtual-reality augmented exposure (i.e. olfactory stimulation, heart rate, and skin conductance); group therapy to address sleep, anger, depression, and social isolation; homework assignments; and programmed practice. In the 3-week treatment program, each participant receives virtual-reality assisted exposure in the morning followed by in vivo exposure and group therapy (SER) each afternoon for a total of 29 sessions.
  Interventions: Behavioral: Exposure Therapy
- Prolonged Exposure (Active Comparator): 2. Standard Prolonged Exposure (PE; Foa, Hembree, & Rothbaum, 2007) consists of psychoeducation, imaginal exposure to trauma memories, in vivo exposure to situations that are avoided due to their association with the trauma, and emotional processing. The standard protocol consists of 12 imaginal exposure sessions, along with in vivo exposure/homework assignments and listening to a recording of the imaginal sessions at home during the evening.
  Interventions: Behavioral: Exposure Therapy
- Compressed Prolonged Exposure (Active Comparator): 3. Compressed PE consists of 10 standard PE sessions delivered on consecutive work days. The imaginal exposure sessions take place in the morning, with in vivo exposures assigned (not therapist accompanied) for the afternoons. Patients are instructed to listen to the recordings of the imaginal exposure each night. Being most concerned with having enough time for in vivo practice, Session 1 does not start on a Monday, allowing for two full weekends in order to maximize in vivo exposures. Both versions of PE average 36 total treatment hours.
  Interventions: Behavioral: Exposure Therapy

INTERVENTIONS:
Behavioral: Exposure Therapy — Exposure Therapy is used to reduce the symptoms of PTSD

SUMMARY:
The purpose of this requirement is to identify an effective exposure psychotherapy paradigm for the treatment of Post-Traumatic Stress Disorder (PTSD) in active duty service members and veterans by comparing different exposure psychotherapy modalities. The long-term goal of exposure psychotherapy is to improve the mental health of U.S. service members and veterans with military-related PTSD. Recovery from PTSD will reduce the economic burden not only for those persons experiencing PTSD, but also for the health care system and society as a whole (Galovski & Lyons, 2004).

DETAILED DESCRIPTION:
This study will provide an evaluation of performance and suitability of the compressed versions of exposure psychotherapy to support the capability gap for the treatment of active duty service members and veterans with PTSD by comparing different exposure psychotherapy modalities. The overall objective of this study is to determine if compressed psychotherapy can be used as an effective alternative treatment for PTSD and to compare the impact of TMT and PE on social, familial, and occupational impairment. The primary objectives will be to compare 1) 3 week TMT with 12 week PE and 2) 3 week TMT with 2 week PE for the effectiveness of reducing PTSD symptoms in a gated approach or some other method to control for multiplicity. Outcomes will be determined based upon self-report, clinician ratings, as well as other aspects of psychopathology, and social/emotional functioning. The addition of the TMT group component will be assessed in particular to determine its impact on social, familial, and occupational impairment. Blood samples should be collected from participants at baseline and at the end of the treatment period in order to identify PTSD biomarkers, e.g. predictors of response, biological subtypes of PTSD, and therapeutic markers. Collection, storage, and transfer of the blood samples to DoD should be performed according to standardized protocols provided by the DoD. One or more site visits may occur in order to assess adherence to standardized protocols.

ELIGIBILITY:
Inclusion Criteria:

* Active duty military personnel with a diagnoses of PTSD
* Traumatic event must have occurred during military service
* Military sexual trauma limited to attempted or completed sexual assault.

Exclusion Criteria:

* Acute cardiac difficulties
* Severe comorbid substance use disorders.
* Diagnosis of schizophrenia or other psychotic disorders
* Diagnosis of antisocial personality disorder
* Moderate or severe traumatic brain injury (TBI)
* Use of benzodiazepines

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on the Clinician-Administered PTSD Scale for DSM-5 | 1 week posttreatment
  PTSD symptoms rating scale (severity and frequency) administered by blinded clinician
Change from Baseline on the Clinician-Administered PTSD Scale for DSM-5 | 3 months posttreatment
  PTSD symptoms rating scale (severity and frequency) administered by blinded clinician
Change from Baseline on the Clinician-Administered PTSD Scale for DSM-5 | 6 months posttreatment
  PTSD symptoms rating scale (severity and frequency) administered by blinded clinician

SECONDARY OUTCOMES:
Change from Baseline on the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | 1 week posttreatment
  Patient Self Report of PTSD symptoms
Change from Baseline on the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | 3 months posttreatment
  Patient Self Report of PTSD symptoms
Change from Baseline on the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | 6 months posttreatment
  Patient Self Report of PTSD symptoms
Change from Baseline on the Traumatic Life Events Questionnaire (TLEQ) | 1 week posttreatment
  self-report measure assessing lifetime history of 22 traumatic events
Change from Baseline on the Traumatic Life Events Questionnaire (TLEQ) | 3 months posttreatment
  self-report measure assessing lifetime history of 22 traumatic events
Change from Baseline on the Traumatic Life Events Questionnaire (TLEQ) | 6 months posttreatment
  self-report measure assessing lifetime history of 22 traumatic events
Change from Baseline on the Trauma-Related Guilt Inventory (TRGI) | 1 week posttreatment
  32-item measure rating 3 domains of trauma-related guilt cognitions (Global Guilt, Distress, and Guilt Cognitions)
Change from Baseline on the Trauma-Related Guilt Inventory (TRGI) | 3 months posttreatment
  32-item measure rating 3 domains of trauma-related guilt cognitions (Global Guilt, Distress, and Guilt Cognitions)
Change from Baseline on the Trauma-Related Guilt Inventory (TRGI) | 6 months posttreatment
  32-item measure rating 3 domains of trauma-related guilt cognitions (Global Guilt, Distress, and Guilt Cognitions)
Change from Baseline on the Posttraumatic Cognitions Inventory (PTCI) | 1 week posttreatment
  36-item measure assessing 3 domains of trauma-related cognitions (Negative Cognitions about Self, Negative Cognitions about the World, and Self-Blame)
Change from Baseline on the Posttraumatic Cognitions Inventory (PTCI) | 3 months posttreatment
  36-item measure assessing 3 domains of trauma-related cognitions (Negative Cognitions about Self, Negative Cognitions about the World, and Self-Blame)
Change from Baseline on the Posttraumatic Cognitions Inventory (PTCI) | 6 months posttreatment
  36-item measure assessing 3 domains of trauma-related cognitions (Negative Cognitions about Self, Negative Cognitions about the World, and Self-Blame)
Change from Baseline on the Moral Injury Event Scale (MIES) | 1 week posttreatment
  patient-report measure assessing psychological distress associated with violations of moral standards.
Change from Baseline on the Moral Injury Event Scale (MIES) | 3 months posttreatment
  patient-report measure assessing psychological distress associated with violations of moral standards.
Change from Baseline on the Moral Injury Event Scale (MIES) | 6 months posttreatment
  patient-report measure assessing psychological distress associated with violations of moral standards.
Change from baseline on the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | 1 week posttreatment
  patient report of impairment in six domains: cognition, mobility, self-care, getting along with people, life activities (at home and work), and participation in society
Change from baseline on the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | 3 months posttreatment
  patient report of impairment in six domains: cognition, mobility, self-care, getting along with people, life activities (at home and work), and participation in society
Change from baseline on the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | 6 months posttreatment
  patient report of impairment in six domains: cognition, mobility, self-care, getting along with people, life activities (at home and work), and participation in society
Change from baseline on the Quality of Life Scale (QOLS) | 1 week posttreatment
  Patient report of 6 domains of life: independence, recreation, personal development and fulfillment, material and physical well-being, relationships with others, and community and civic involvement
Change from baseline on the Quality of Life Scale (QOLS) | 3 months posttreatment
  Patient report of 6 domains of life: independence, recreation, personal development and fulfillment, material and physical well-being, relationships with others, and community and civic involvement
Change from baseline on the Quality of Life Scale (QOLS) | 6 months posttreatment
  Patient report of 6 domains of life: independence, recreation, personal development and fulfillment, material and physical well-being, relationships with others, and community and civic involvement
Change from baseline on the Connor-Davidson Resilience Scale (CD-RISC) | 1 week posttreatment
  Patient report of coping ability
Change from baseline on the Connor-Davidson Resilience Scale (CD-RISC) | 3 months posttreatment
  Patient report of coping ability
Change from baseline on the Connor-Davidson Resilience Scale (CD-RISC) | 6 months posttreatment
  Patient report of coping ability
Change from baseline on the Patient Health Questionnaire-9 (PHQ-9) | 1 week posttreatment
  Patient report measure of depression symptoms
Change from baseline on the Patient Health Questionnaire-9 (PHQ-9) | 3 months posttreatment
  Patient report measure of depression symptoms
Change from baseline on the Patient Health Questionnaire-9 (PHQ-9) | 6 months posttreatment
  Patient report measure of depression symptoms
Change from baseline on the Generalized Anxiety Disorder-7 (GAD-7) | 1 week posttreatment
  Patient report measure of general anxiety symptoms
Change from baseline on the Generalized Anxiety Disorder-7 (GAD-7) | 3 months posttreatment
  Patient report measure of general anxiety symptoms
Change from baseline on the Generalized Anxiety Disorder-7 (GAD-7) | 6 months posttreatment
  Patient report measure of general anxiety symptoms
Change from baseline on the Dimensions of Anger Reactions-5 (DAR-5) | 1 week posttreatment
  Patient report measure of anger
Change from baseline on the Dimensions of Anger Reactions-5 (DAR-5) | 3 months posttreatment
  Patient report measure of anger
Change from baseline on the Dimensions of Anger Reactions-5 (DAR-5) | 6 months posttreatment
  Patient report measure of anger
Change from baseline on the Clinical Global Impressions Scales (CGI) | 1 week posttreatment
  Clinician rated scales to evaluate the severity of pretreatment psychopathology and treatment change
Change from baseline on the Clinical Global Impressions Scales (CGI) | 3 months posttreatment
  Clinician rated scales to evaluate the severity of pretreatment psychopathology and treatment change
Change from baseline on the Clinical Global Impressions Scales (CGI) | 6 months posttreatment
  Clinician rated scales to evaluate the severity of pretreatment psychopathology and treatment change
Sleep actigraphy - change from baseline in total sleep time | 1 week posttreatment
  Objective assessment of sleep
Sleep actigraphy - change from baseline in total sleep time | 3 months posttreatment
  Objective assessment of sleep
Sleep actigraphy - change from baseline in total sleep time | 6 months posttreatment
  Objective assessment of sleep
Sleep actigraphy - change from baseline in sleep onset latency | 1 week posttreatment
  Objective assessment of sleep (# of minutes to sleep onset after getting into bed)
Sleep actigraphy - change from baseline in sleep onset latency | 3 months posttreatment
  Objective assessment of sleep (# of minutes to sleep onset after getting into bed)
Sleep actigraphy - change from baseline in sleep onset latency | 6 months posttreatment
  Objective assessment of sleep (# of minutes to sleep onset after getting into bed)
Sleep actigraphy - change from baseline in sleep efficiency | 1 week posttreatment
  Objective assessment of sleep (% of time in bed spent sleeping)
Sleep actigraphy - change from baseline in sleep efficiency | 3 months posttreatment
  Objective assessment of sleep (% of time in bed spent sleeping)
Sleep actigraphy - change from baseline in sleep efficiency | 6 months posttreatment
  Objective assessment of sleep (% of time in bed spent sleeping)
Sleep actigraphy - change from baseline in wake minutes after sleep onset | 1 week posttreatment
  Objective assessment of sleep (# of minutes awake after falling asleep)
Sleep actigraphy - change from baseline in wake minutes after sleep onset | 3 months posttreatment
  Objective assessment of sleep (# of minutes awake after falling asleep)
Sleep actigraphy - change from baseline in wake minutes after sleep onset | 6 months posttreatment
  Objective assessment of sleep (# of minutes awake after falling asleep)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Beidel, Ph.D., Principal Investigator — University of Central Florida
Locations (1):
- UCF RESTORES, University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No